CLINICAL TRIAL: NCT05866978
Title: An Integrated Approach to Health, Wellbeing, and Productivity at Work
Acronym: ITASPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R22A547; SJ-927 (Other: Ethics Committee in Region Zealand, Denmark); REG-034-2021 (Other: The Danish data protection agency)
Record Dates: First submitted 2023-03-29; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Musculoskeletal Disorder; Mental Health Issue; Work-related Illness; Safety Issues; Work Environment Adverse Effects
Keywords: total worker health; occupational safety and health; intervention development; cleaning assistants; pain and injury; wellbeing; working conditions; work environment; workhealth improvement network
MeSH Terms: conditions — Musculoskeletal Diseases; Occupational Stress; Pain; Wounds and Injuries | interventions — Health

STUDY DESIGN:
Intervention Model Description: Using a stepped-wedge design, participants at the enrolled worksites function as their own control. Thus, the effect of the intervention is evaluated as in an RCT design. All employees are asked to complete a short screening questionnaire. Those who wish to participate are invited to the data collection containing: Signing of consent, measurements of height, body weight, fat percentage and blood pressure and answering a questionnaire. No preparation is required of the participants before data collection begins. All intervention activities and health checks take place at the participants' workplace during paid working hours. Calculation, analysis and interpretation of data will take place at the Department of Occupational and Social Medicine, Holbæk Hospital.
  The intervention activities are developed by a local commitee including participants and managers, acoording a participatory approach and following the Work Health Improvements Network concept.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An integrated workplace intervention (Other): Intervention: A group of employees at each workplace will develop and implement their own project activities at meetings four times during the intervention. Activities are implemented at workplaces for all employees. Employees will participate in one screening questionnaire prior to the intervention followed by five health checks and interview based questionnaires.
  Interventions: Behavioral: Integrated Approach to Health, Wellbeing, and Productivity at Work (ITASPA)
- Reference (No Intervention): Reference: No intervention activities.

INTERVENTIONS:
Behavioral: Integrated Approach to Health, Wellbeing, and Productivity at Work (ITASPA) — The intervention investigates the effect of the Australian WorkHealth Improvement Network (WIN) program and the Total Worker Health (TWH) concepts in a Danish context among blue-collar workers.
  Arms: An integrated workplace intervention

SUMMARY:
The goal of the workplace intervention study 'An Integrated Approach to Health, Wellbeing, and Productivity at Work (ITASPA)' is to examine the effect of the Australian WorkHealth Improvement Network (WIN) program in a Danish context among blue-collar workers. The project is evaluated via its effect on: 1) Musculoskeletal disorders (MSD), 2) Functionality, 3) Psychosocial wellbeing, and 4) Safety culture. Based on identified work health challenges at the included workplace, a group of employees at each worksite will develop and implement their own health promoting activities. Remaining employees will participate in one screening questionnaire prior to the intervention followed by five health checks and interview based questionnaires. All intervention activities and health checks take place at the participants' workplace during paid working hours. In our study design, participants will be compared to themselves and their previous measurements. Furthermore, we will compare the worksites.

DETAILED DESCRIPTION:
The aim of the 'Integrated Approach to Health, Wellbeing, and Productivity at Work (ITASPA)' project is to investigate the effect of the Australian WorkHealth Improvement Network (WIN) program and the Total Worker Health (TWH) concepts in a Danish context among blue-collar workers. The project is evaluated via its effect on: 1) Musculoskeletal disorders (MSD), 2) Functionality, 3) Psychosocial wellbeing, and 4) Safety culture. In addition, we evaluate the intervention effect on BMI, heart rate, and blood pressure. Furthermore, the ITASPA project aims to examine the degree of implementation of the initiated initiatives and identify barriers and facilitating factors for implementation. This contributes to the knowledge about what characterizes best practices for the implementation of integrated workplace interventions.

Based on identified work health challenges at the included worksites, a group of employees at each workplace will develop and implement their own project activities. Remaining employees will participate in one screening questionnaire prior to the intervention followed by five health checks and interview based questionnaires. All intervention activities and health checks take place at the participants' workplace during paid working hours.

ITASPA is a workplace intervention, conducted in a stepped wedge design. The stepped wedge design are assumed to increase the willingness to participate as it allows all workers to receive the intervention. The workers function as their own control and thereby, the stepped wedge design allows for an effect-evaluation, mimicking an RCT design.

To increase the transferring of the WIN program to a broad variety of Danish worksites, both public and private worksites are aimed to be enrolled. The worksites will be enrolled on basis of their willingness to perform the ITASPA activities during paid worktime and participation in the scientific evaluation of the ITASPA project.

The ITASPA project will be organized by a steering group consisting of the ITASPA project managers, representatives from the senior management at the enrolled worksites, and the ITASPA facilitators from the Department of Occupational and Social Medicine at Holbæk Hospital, Denmark. Moreover, the steering group includes an advisory board consisting of the developers of the WIN program and TWH concept. The advisory board will provide information about international experiences with integrated workplace interventions to assist the development of workplace health interventions in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Employed at one of the enrolled worksites ≥ 20 hours/week, providing an informed signed consent prior to participation.

Exclusion Criteria:

* Being pregnant; not being able to understand and speak Danish or English

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of musculoskeletal disorders from baseline to 6, 9, 12 and 15 months after randomization | Data on musculoskeletal disorders are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  The Short Form of the Örebro Musculoskeletal Pain Screening Questionnaire will be used to measure musculoskeletal disorders
Change of functionality from baseline to 6, 9, 12 and 15 months after randomization | Data on functionality are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Functionality will be measured by the ICF-based Work Rehabilitation Questionnaire (WORQ) (https://myworq.org/)
Change of psychosocial wellbeing from baseline to 6, 9, 12 and 15 months after randomization | Data on psychosocial wellbeing are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Psychosocial wellbeing will be measured via the Health Survey SF-12
Change of safety culture from baseline to 6, 9, 12 and 15 months after randomization | Data on safety culture are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Safety culture will be measured by the Nordic Occupational Safety Climate Questionnaire (NOSACQ-50)
Change of body weight (kg) from baseline to 6, 9, 12 and 15 months after randomization | Data on body weight (kg) are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Bodyweight will be measured while the participant is wearing light clothes and no shoes. The estimated weight of clothes (1.5 kg) will be subtracted from body weight. Percent body fat will be estimated by bioelectric-impedance-analysis. Both body weight and percent body fat will be measured by a Segmental Body Composition Monitor, Innerscan V, BC545N (TANITA, produced in Japan). If participants have a pacemaker or are pregnant, the analysis of percent body fat will not be made. Body height will be measured on a mobile stadiometer Seca 213 (Seca, produced in China). Body mass index (BMI) will be estimated by the equation of BMI = (body weight (kg)/body height (m)2).
Change of percent body fat from baseline to 6, 9, 12 and 15 months after randomization | Data on percent body fat are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Percent body fat will be measured while the participant is wearing light clothes and no shoes. The estimated weight of clothes (1.5 kg) will be subtracted from body weight. Percent body fat will be estimated by bioelectric-impedance-analysis. Both body weight and percent body fat will be measured by a Segmental Body Composition Monitor, Innerscan V, BC545N (TANITA, produced in Japan). If participants have a pacemaker or are pregnant, the analysis of percent body fat will not be made. Body height will be measured on a mobile stadiometer Seca 213 (Seca, produced in China). Body mass index (BMI) will be estimated by the equation of BMI = (body weight (kg)/body height (m)2).
Change of resting heart rate (beats per minute) from baseline to 6, 9, 12 and 15 months after randomization. | Data on heart rate are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Resting heart rate will be measured three times on the left arm after 15 minutes of sitting at rest using an Omron Model M3, automatic upper arm BP monitor (Omron healthcare, produced in Vietnam).
Change of blood pressure (mmHg) from baseline to 6, 9, 12 and 15 months after randomization. | Blood pressure are collected 3 months after randomization. Additional follow up data are collected 6, 9, 12 and 15 months after randomization.
  Blood pressure will be measured three times on the left arm after 15 minutes of sitting at rest using an Omron Model M3, automatic upper arm BP monitor (Omron healthcare, produced in Vietnam).

SECONDARY OUTCOMES:
Change of sickness absence from 12 months prior to the randomization and 12 months after the last (15 months) follow up. | Data on sickness absence are collected from 12 months prior to the randomization and 12 months after the last (15 months) follow up.
  Information on sickness absence is provided by the administration at workplaces

CONTACTS AND LOCATIONS:
Overall Officials: Mette Korshøj, PhD, Principal Investigator — Holbaek Hospital
Locations (1):
- Department of Occupational and Social Medicine, Holbæk, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korshoj M, Poulsen VR, Skold MB, Autrup SK, Oldenburg B, Mortensen OS. An integrated approach to health, wellbeing, and productivity at work: a design of a stepped wedge worksite intervention study. BMC Public Health. 2023 Jun 2;23(1):1057. doi: 10.1186/s12889-023-16014-x. PMID 37268907